CLINICAL TRIAL: NCT00057954
Title: A Phase II Study of Reduced Intensity Allogeneic Bone Marrow Transplantation for the Treatment of Relapsed Non-Hodgkin and Hodgkin Lymphoma
Brief Title: Reduced-Intensity Regimen Before Allogeneic Transplant for Patients With Relapsed Non-Hodgkin's or Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000285659; U10CA021115 (NIH); E1402 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Photopheresis; Pentostatin; Whole-Body Irradiation; Radiotherapy; Cyclosporine; Cyclosporins; Mycophenolic Acid; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transplant (Experimental): Reduced toxicity conditioning regimen followed by allogeneic sibling or unrelated transplant. The conditioning regimen includes Extracorporeal Photopheresis, Pentostatin and total body irradiation (TBI). After allogeneic bone marrow transplantation, cyclosporin, mycophenolate mofetil (MMF), and methotrexate (MTX) will be given to prevent graft-versus-host disease (GVHD).
  Interventions: Procedure: Extracorporeal Photopheresis; Drug: Pentostatin; Radiation: Total body irradiation (TBI); Procedure: Allogeneic bone marrow transplantation; Drug: Cyclosporin (CSA); Drug: Mycophenolate mofetil (MMF); Drug: Methotrexate (MTX)

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis — Day -7 to -4: Extracorporeal Photopheresis may be given as an outpatient therapy on two consecutive days any time between days -7 to -4. This must be performed on UVAR or XTS photopheresis machines (Therakos, Inc.) according to standard procedure as per manufacturer's guidelines.
  Other Names: extracorporeal photochemotherapy
Drug: Pentostatin — Day -3, -2: Pentostatin 4 mg/m²/d by continuous IV infusion (Total dose = 8 mg/m²)
  Other Names: DCF,; 2-Deoxycoformycin,; Nipent
Radiation: Total body irradiation (TBI) — Day -1: TBI 400 cGy total dose given in two 200cGy doses. Patients who have received TBI for a previous transplant or radiation as part of previous treatment for a lymphoid malignancy will receive only 200 cGy in 1 dose.
  Other Names: radiation therapy
Procedure: Allogeneic bone marrow transplantation — Day 0: Infusion of unmanipulated allogeneic bone marrow or stem cells. Minimum cell dose of 2 x 106 CD34 cells/kg recipient and no more than 10 x 10^6 CD34/kg
  Other Names: allogeneic stem cell transplantation
Drug: Cyclosporin (CSA) — Cyclosporin A or tacrolimus will be administered according to institutional GVHD prophylaxis protocols. Therapeutic levels will be maintained and patients will be switched to oral agents when they can tolerate
  Other Names: Sandimmune,; cyclosporin A,; CSA,; Neoral,; Gengraf
Drug: Mycophenolate mofetil (MMF) — At day 100 MMF will be introduced at a dose of 250 mg po BID and cyclosporine or tacrolimus will be tapered according to the discretion of the investigator. The dosage will be escalated to a maximum of 2 g/d at the discretion of the attending physician and will be tapered and discontinued at 12 months if there is no active cGVHD. Doses should be given on an empty stomach
  Other Names: Cellcept,; mycophenolic acid,; Lilly-68618,; RS-61443,; MMF
Drug: Methotrexate (MTX) — The dose of Methotrexate is based on the corrected ideal body weight for patients with > 33% above ideal weight.
  Day +1 MTX 15 mg/m² IV push; Day +3 MTX 10 mg/m² IV push (May be omitted if patient develops mouth sores.)
  Other Names: Methotrexate sodium,; MTX,; Mexate,; Mexate-AQ,; Folex,; Folex PFS,; Abitrexate,; Rheumatrex,; Amethopterin

SUMMARY:
RATIONALE: Photopheresis allows patient white blood cells to be treated with ultraviolet (UV) light and drugs outside the body to inactivate T cells. Pentostatin may suppress the immune system and reduce the chance of developing graft-versus-host disease (GVHD) following bone marrow transplantation. Combining photopheresis with pentostatin and total-body irradiation may be effective in killing cancer cells before bone marrow transplantation.

PURPOSE: This phase II trial is studying how well giving photophoresis together with pentostatin and total-body irradiation as a reduced-intensity regimen before allogeneic bone marrow transplantation works in treating patients with relapsed non-Hodgkin's or Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rate of stable engraftment of donor cells in patients with relapsed non-Hodgkin's or Hodgkin's lymphoma treated with a reduced toxicity conditioning regimen followed by allogeneic (sibling or unrelated) bone marrow transplantation.
* Determine the extent and duration of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the 100-day overall survival and long-term progression-free survival of patients treated with this regimen.
* Evaluate the feasibility of collection of molecular chimerism studies at baseline, days 30, 100, 6 months and one and two years and at relapse.

OUTLINE: This is a multicenter study.

* Conditioning regimen: Patients undergo extracorporeal photopheresis using methoxsalen and UV light on 2 consecutive days between days -7 to -4. Patients receive pentostatin intravenously (IV) continuously on days -3 to -2 and undergo total body irradiation on day -1.
* Allogeneic bone marrow transplantation: Patients undergo infusion of allogeneic bone marrow or stem cells on day 0.
* Graft-versus-host disease prophylaxis: Patients receive oral or IV cyclosporine beginning on day -1 and continuing until 6 months after transplantation, oral mycofenolate mofetil beginning on day 100 and continuing for 1 year, and methotrexate IV on days 1 and 3.

Patients are followed at day 100, every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 1.8 years.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hodgkin's or Hodgkin's lymphoma that has relapsed following either a course of high dose chemotherapy or autologous stem cell transplantation.
* >= 90 days from prior transplant.
* Have a suitable human leukocyte antigen (HLA)-matched related bone marrow donor or a compatible matched unrelated bone marrow donor by molecular typing at HLA A, B, C, D, DR.
* Physically and psychologically capable of undergoing bone marrow transplantation and its attendant period of strict isolation.
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Be able to receive 400 cGy Total Body Irradiation (TBI).
* Pulmonary function tests: Diffusing capacity or Transfer factor of the lung for carbon monoxide (DLCO) >= 50% predicted, the forced expiratory volume in 1 second (FEV1) >= 50% predicted.
* Left ventricular ejection fraction (LVEF) at least 45% by Multi Gated Acquisition Scan (MUGA) or echocardiogram.
* Renal function: creatinine clearance > 50 ml/min.
* Liver function tests: < 3 x Upper Limit of Normal (ULN). Liver function test include serum glutamic oxaloacetic transaminase (SGOT) (Aspartate transaminase (AST)), Serum Glutamic Pyruvate Transaminase (SGPT) (Alanine transaminase (ALT)), and bilirubin.

Exclusion Criteria:

* Human immunodeficiency virus positive (HIV+) patients (test positive for P21 antibodies to HIV).
* Evidence of active infection (have received parenteral antibiotics <= 2 weeks prior to registration).
* Pregnant or breast-feeding women.
* Curable with any other therapeutic interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-11-09 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine M. Foss, MD, Study Chair — Yale University
Locations (19):
- United States (19):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between June 1, 2005 and October 10, 2007 with the first patient accrued on November 9, 2005.
Groups:
- Transplant: Reduced toxicity conditioning regimen followed by allogeneic (sibling or unrelated) transplant.
Period: Overall Study
Arm/Group | Transplant
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Transplant: Reduced toxicity conditioning regimen followed by allogeneic sibling or unrelated transplant.
Arm/Group | Transplant
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 47 [21 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Successful Engraftment
Time Frame: Assessed daily during inpatient stay
Population: all enrolled 6 patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Transplant
Number analyzed (Participants) | 6
Proportion of participants | 1 [0.5 to 1.0]

2. Secondary Outcome: 100-day Overall Survival
Description: Proportion of patients who survived 100 days or more after enrolled on the study
Time Frame: Assessed at least twice a week for the first 60 days and weekly until day 100.
Population: all 6 enrolled patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Transplant
Number analyzed (Participants) | 6
Proportion of participants | 0.83 [0.54 to 1.0]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as time from enrollment to disease progression or death from any cause, whichever occurred first. Patients who did not have progression-free survival events were censored at last date of disease assessment.
Time Frame: Assessed day 100 post transplant and every 3 months during year 1, every 6 months during years 2-3, then every 12 months during years 4-5 or through diagnosis of disease progression
Population: all 6 enrolled patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Transplant
Number analyzed (Participants) | 6
days | 104 [66 to NA] — upper limit of confidence interval (CI) has not been reached

ADVERSE EVENTS:
Time Frame: Assessed every 30 days while on treatment and for 30 days after the end of treatment.
Arm/Group | Transplant
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant (N=6)
Anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Leukocytes, decreased) (Investigations) | 6
Lymphopenia (Investigations) | 6
Neutropenia (Neutrophils, decreased) (Investigations) | 6
Thrombocytopenia (Platelets, decreased) (Investigations) | 4
Fatigue (General disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 2
Head/headache (Nervous system disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant (N=6)
Anemia (Blood and lymphatic system disorders) | 6
Leukopenia (Leukocytes, decreased) (Investigations) | 6
Lymphopenia (Investigations) | 5
Neutropenia (Neutrophils, decreased) (Investigations) | 5
Thrombocytopenia (Platelets, decreased) (Investigations) | 6
Fatigue (General disorders) | 1
Fever w/o neutropenia (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
GI-other (Gastrointestinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 6
Creatinine, increased (Investigations) | 5
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No